CLINICAL TRIAL: NCT06864507
Title: A Randomized, Double-blind, Placebo-controlled Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HS-10561 Capsule in Healthy Chinese Adults and Patients With Chronic Spontaneous Urticaria.
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HS-10561 Capsule in Healthy Chinese Adults and Patients With Chronic Spontaneous Urticaria.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10561-101
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Chronic spontaneous urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HS-10561 Dose 1 (Experimental): HS-10561, Dose 1
  Interventions: Drug: HS-10561
- HS-10561 Dose 2 (Experimental): HS-10561, Dose 2
  Interventions: Drug: HS-10561
- HS-10561 Dose 3 (Experimental): HS-10561, Dose 3
  Interventions: Drug: HS-10561
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10561 — Single and multiple doses of HS-10561 orally
  Arms: HS-10561 Dose 1; HS-10561 Dose 2; HS-10561 Dose 3
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 1/2 clinical study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of HS-10561 capsule in healthy Chinese adults and patients with chronic spontaneous urticaria.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.(SD)
* Healthy adults aged 18-45 years (inclusive) at the time of signing the informed consent form;(SD)
* Male participants weighing ≥ 50 kg and female participants weighing ≥ 40 kg; body mass index (weight/square of height (kg/m2)) within the range of 18-30 kg/m2 (inclusive);(SD)
* Female participants and male participants (including their female partners) agree to use highly effective methods of contraception from the date of signing the informed consent form until 30 days after the last dose;(SD)
* Without history of severe respiratory, gastrointestinal (such as inflammatory bowel disease, Crohn's disease, chronic diarrhea, etc.), neurological, circulatory, urinary, endocrine, musculoskeletal, immune system disorders, or a history of tumors prior to screening.(SD)
* Written informed consent must be obtained before any assessment is performed.(MD and Phase 2)
* Healthy adults aged 18-65 years (inclusive) at the time of signing the informed consent form;(MD and Phase 2)
* Have been diagnosed with chronic spontaneous urticaria for ≥6 months at the time of screening;(MD and Phase 2)
* Female participants and male participants (including their female partners) agree to use highly effective methods of contraception from the date of signing the informed consent form until 30 days after the last dose.(MD and Phase 2)

Exclusion Criteria:

* Have clinically significant abnormalities in vital signs, physical examination, laboratory tests, chest X-ray/CT, or abdominal ultrasound during the screening period, which, as assessed by the investigator, may increase the participants' risk or affect the scientific validity of the study;(SD)
* Females with a positive blood pregnancy test, breastfeeding females, or participants planning to become pregnant during the study period;(SD)
* Any physiological or psychological condition or disease, as determined by the investigator, that could increase the risk, affect the participants' compliance, or impact the participants' ability to complete the study.(SD)
* Chronic urticaria with a clear primary or sole trigger (chronic inducible urticaria);(MD and Phase 2)
* Clearly defined predominant or sole trigger of their chronic urticaria (chronic inducible urticaria);(MD and Phase 2)
* Other diseases with symptoms of urticaria or angioedema;(MD and Phase 2)
* Other skin disease associated with chronic itching that might influence in the investigators opinion the study evaluations and results;(MD and Phase 2)
* Pregnant or nursing (lactating) women.(MD and Phase 2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-09-27 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation.(Phase 1) | SD：up to 7 days，MD：up to 35 days
  Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation.
Change from baseline in Weekly Urticaria Activity Score (UAS7) at Week 4 (Phase 2) | Week 4
  The Weekly Urticaria Activity Score (UAS7) is a simple scoring system to evaluate urticaria signs and symptoms. It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42 (highest urticaria severity), and a minimum possible score of 0.

SECONDARY OUTCOMES:
Cmax | Day 1 up to Day 4 (SD), Day 1 up to Day 35 (MD)
  Maximum plasma concentration
Tmax | Day 1 up to Day 4 (SD), Day 1 up to Day 35 (MD)
  Time to reach Cmax
AUC | Day 1 up to Day 4 (SD), Day 1 up to Day 35 (MD)
  Area under the plasma concentration-time curve
t½ | Day 1 up to Day 4 (SD), Day 1 up to Day 35 (MD)
  Terminal half-life
CL/F | Day 1 up to Day 4 (SD), Day 1 up to Day 35 (MD)
  Apparent clearance
Vd/F | Day 1 up to Day 4 (SD), Day 1 up to Day 35 (MD)
  Apparent volume of distribution
Rac | Day 1 up to Day 4 (SD), Day 1 up to Day 35 (MD)
  Accumulation ratio
Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation.(Phase 2) | up to 16 weeks
  Incidence, severity and association with the study drug of adverse events (AEs), serious AEs (SAEs), and AEs leading to discontinuation；Clinically significant changes in physical examination and anamnesis, vital signs, ECG, safety laboratory will be reported under (S)AEs.
Change from baseline in Weekly Itch Severity Score (ISS7) at Week 12(Phase 2) | Week 12
  The severity of the itch was recorded by the participant daily in their electronic Diary, on a scale of 0 (none) to 3 (severe). A weekly score (ISS7) was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 - 21 (highest itch severity).
Change from baseline in Weekly Hives Severity Score (HSS7) at Week 12(Phase 2) | Week 12
  The hives (wheals) severity score, defined by number of hives, was recorded by the participant daily in their electronic Diary, on a scale of 0 (none) to 3 (> 12 hives/12 hours). A weekly score (HSS7) was derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score was therefore 0 - 21 (highest hives activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Hospital of Skin Disease, Shanghai, Shanghai Municipality, China